CLINICAL TRIAL: NCT06208891
Title: Clinical Outcomes of Robotic Myomectomy: Comparisons of Without Versus With Temporary or Permanent Uterine Artery Occlusion.
Brief Title: Clinical Outcomes of Robotic Myomectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 112185-E
Record Dates: First submitted 2023-12-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Women With Uterine Myoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Robotic myomectomy: Women who received robotic myomectomy
  Interventions: Procedure: Robotic myomectomy

INTERVENTIONS:
Procedure: Robotic myomectomy — Robotic assisted laparoscopic myomectomy

SUMMARY:
To identify the predictors of perioperative outcomes in women who receive robotic myomectomy

DETAILED DESCRIPTION:
Uterine myoma is the most common gynecological tumor. Current surgical management was inclusive of conventional abdominal myomectomy, laparoscopy-assisted myomectomy, robotic-assisted myomectomy. The aim of this study was to identify the predictors of perioperative outcomes in women who receive robotic myomectomy

ELIGIBILITY:
Inclusion criteria

* >20 years old women
* women who received robotic myomectomy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women who received robotic myomectomy
Study Population: Women who received robotic-assisted myomectomy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical time | 1 week
  Factors (e.g., the location and largest diameter of the uterine myoma) predicting surgical time

SECONDARY OUTCOMES:
Intraoperative blood loss | 1 week
  Factors (e.g., the location and largest diameter of the uterine myoma) predicting intraoperative blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan